CLINICAL TRIAL: NCT05307146
Title: Study of Brain Activity in Candidates for Epilepsy Surgery
Brief Title: Brain Activity in Epilepsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Tom Theys, Principal Investigator, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: S53126
Record Dates: First submitted 2019-01-18; First posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- micro/macro electrode (Experimental)
  Interventions: Device: macro/micro electrode recording

INTERVENTIONS:
Device: macro/micro electrode recording — intracranial macro/micro-electrode placement at the cerebral cortex or in deeper brain areas with te use of macro/micro electrode recording. Macro/micro electrodes are placed at the cerebral cortex or in deeper brain areas in order to precisely identify the epileptogenic focus

SUMMARY:
Prospective interventional study with implantation of micro-electrodes to study the brain networks in epilepsy at high spatiotemporal resolution.

DETAILED DESCRIPTION:
The goal of this trial is to study brain activity in epilepsy at high spatiotemporal resolution. Apart from the epileptogenic network (dysfunctional areas), the investigators will study human brain function.

The use of micro-electrode arrays allows to study the human brain a high spatiotemporal resolution, even at the single neuron level.

Scientific objectives of the current project:

* To record neural signals from macro-electrodes and delineate the epileptogenic network and study brain function during specific tasks.
* To record neural signals from micro-electrodes and delineate the epileptogenic network and study brain function during specific tasks.
* Identifying pivotal regions for BMI applications and developing online decoding algorithms.
* Comparing neural recordings to fMRI activity

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 yo
* Epilepsy patients undergoing intracranial electrode placement.
* Able to understand the procedure involved and to consent.

Exclusion Criteria:

* Age < 18 yo
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-12-18 (Actual); Primary Completion 2035-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Electrophysiological recordings: single neuron recordings | 15 years
  The investigators will investigate the epileptogenic network by recording neural activity at different spatiotemporal scales and using different modalities. The investigators will be looking at * Electrophysiological recordings:
  - single neuron recordings (outcome measure: spike rate)
Electrophysiological recordings: LFP | 15 years
  The investigators will investigate the epileptogenic network by recording neural activity at different spatiotemporal scales and using different modalities. The investigators will be looking at * Electrophysiological recordings:
  - local field potentials (LFP) (outcome measure: mainly power in the beta and gamma band, but also alfa and theta band)
fMRI recordings | 15 years
  * fMRI recordings (outcome measure: Blood Oxygen Level Dependent (BOLD) signal increases/decreases)
  By performing electrophysiological recordings and fMRI recordings in the same subjects, we will be able to compare both modalities with each other.

SECONDARY OUTCOMES:
Neurophysiological study of different brain areas: power gamma band | 15 years
  Since electrodes are placed for clinical purposes, the investigators will also use these electrodes to investigate normal neural functions of the human brain: vision, perception and motor.
  * Macro-electrodes record local field potentials (LFP). The main outcome measure for visual research is the power in the gamma band. The main outcome measure for motor research is power increase in the beta and gamma band.
Neurophysiological study of different brain areas: spike activity | 15 years
  * Micro-electrodes and multi-electrode arrays (Utah-array) record local field potentials (LFP) and spike-activity. The outcome measure for spike activity is spike rate. For the local field potentials, the main outcome measure for visual research is the power in the gamma band. The main outcome measure for motor research is power increase in the beta and gamma band.
Neurophysiological study of different brain areas: fMRI | 15 years
  The outcome measure is blood oxygen level dependent (BOLD) signal changed in response to visual and/ or motor experiments.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium